CLINICAL TRIAL: NCT00729651
Title: A Prospective, Randomized, Open-label, Active-controlled Study to Evaluate the Efficacy and Safety of Fosamax Plus D in Postmenopausal Osteoporotic Women
Brief Title: Efficacy and Safety Study of Fosamax Plus D in Postmenopausal Women With Osteoporosis (0217A-263)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0217A-263; MK0217A-263; 2008_015
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Results first posted 2010-04-02 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Alendronate; Cholecalciferol; Fumigant 93

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Alendronate sodium/Cholecalciferol
  Interventions: Drug: alendronate sodium (+) cholecalciferol; Dietary Supplement: Comparator: Calcium
- 2 (Active Comparator): Alendronate sodium
  Interventions: Drug: Comparator: Alendronate sodium (Fosamax); Dietary Supplement: Comparator: Calcium

INTERVENTIONS:
Drug: alendronate sodium (+) cholecalciferol — Alendronate sodium/Cholecalciferol; tablet, once weekly, for 16 weeks
  Other Names: Fosamax Plus D
  Arms: 1
Drug: Comparator: Alendronate sodium (Fosamax) — Alendronate sodium; tablet, once weekly, for 16 weeks
  Arms: 2
Dietary Supplement: Comparator: Calcium — 500 mg oral tablet calcium once daily, for 16 weeks

SUMMARY:
To demonstrate the efficacy/safety of Fosamax Plus D

ELIGIBILITY:
Inclusion Criteria:

* Patient agrees to apply sunscreen and limit sunlight-exposure to 1 hour per day during the study
* Patient has been diagnosed with osteoporosis
* Patient has been postmenopausal for more than 6 months
* Patient has no contraindication to taking oral bisphosphonates
* Patient is eligible for dual energy x-ray absorptiometry in spine or hip

Exclusion Criteria:

* Patients with esophageal dysfunction
* Patients who can not sit or stand at least 30 minutes
* Patients who had a malignant disease or active systemic disease 5 years prior to participating in this trial
* Patients with diseases of bone or mineral metabolism besides osteoporosis or receiving therapies which affect bone metabolism or calcium metabolism
* Patients with history of major gastrointestinal disease (peptic ulcer, malabsorption, esophageal disease, gastritis, gastroduodenitis, etc.) within the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2008-03-20 (Actual); Primary Completion 2009-04-10 (Actual); Study Completion 2009-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim KJ, Min YK, Koh JM, Chung YS, Kim KM, Byun DW, Kim IJ, Kim M, Kim SS, Min KW, Han KO, Park HM, Shin CS, Choi SH, Park JS, Chung DJ, Mok JO, Baek HS, Moon SH, Kim YS, Lim SK; VALUE study group. Efficacy and safety of weekly alendronate plus vitamin D(3) 5600 IU versus weekly alendronate alone in Korean osteoporotic women: 16-week randomized trial. Yonsei Med J. 2014 May;55(3):715-24. doi: 10.3349/ymj.2014.55.3.715. Epub 2014 Apr 1. PMID 24719139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 centers participated in this study (11 - Medical Center of the University, 7 - General Hospital).
  FPE(First patient enrolled) : March-2008, FPI(First patient in) : April-2008, LPO(Last patient out) : April-2009.
Groups:
- Fosamax Plus D: Once weekly Fosamax plus D tablet [Alendronate sodium 70 mg/Cholecalciferol 5600 IU] + once daily calcium formulation [500 mg/day]), 16 weeks
- Fosamax: Once weekly Fosamax 70 mg tablet [Alendronate sodium 70 mg] + once daily calcium formulation [500 mg/day]), 16 weeks
Period: Overall Study
Arm/Group | Fosamax Plus D | Fosamax
Started | 173 | 170
Completed | 154 | 152
Not Completed | 19 | 18
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 5 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 7 | 3
Not completed — Visit 3, 25 OHD level ≤9 ng/mL | 0 | 4
Not completed — Subject's private reason | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fosamax Plus D | Fosamax | Total
Number analyzed (Participants) | 173 | 170 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.59 (7.09) | 65.31 (7.62) | 64.94 (7.36)
Age, Customized [Number; unit: participants]
  <=44 years of age | 0 | 0 | 0
  45-49 years of age | 1 | 0 | 1
  50-59 years of age | 47 | 43 | 90
  60-69 years of age | 85 | 73 | 158
  70-79 years of age | 37 | 51 | 88
  >=80 years of age | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 170 | 343
  Male | 0 | 0 | 0
Patients with/without Vitamin D deficiency [Number; unit: participants] — Vitamin D deficiency means serum 25 OHD (hydroxyvitamin D) below the deficiency level (less than 15 ng/ml) in this study.
  participants
    With Vitamin D deficiency at baseline | 57 | 56 | 113
    Without Vitamin D deficiency at baseline | 116 | 114 | 230
T-score classification by inclusion criteria: A fracture in spine Lumbar 1-4 and T-score ≤ -2.0] [Number; unit: Participants] — T-score: a measurement expressed in standard deviation units from a given mean used in assessment of osteoporosis, equal to a patient's bone mineral density measurement by Dual Energy X-ray Absorptiometry (DEXA) minus the value in a young healthy person, divided by the standard deviation of the measurement in the population.
  Participants
    A fracture in spine Lumbar 1-4 and T-score ≤ -2.0 | 9 | 5 | 14
    Not Applicable | 164 | 165 | 329
T-score classification by inclusion criteria: Femoral neck T-score ≤ -2.5 [Number; unit: Participants] — T-score: a measurement expressed in standard deviation units from a given mean used in assessment of osteoporosis, equal to a patient's bone mineral density measurement by DEXA minus the value in a young healthy person, divided by the standard deviation of the measurement in the population.
  Participants
    Femoral neck T-score ≤ -2.5 | 43 | 58 | 101
    Not Applicable | 130 | 112 | 242
T-score classification by inclusion criteria: Femoral total T-score ≤ -2.5 [Number; unit: Participants] — T-score: a measurement expressed in standard deviation units from a given mean used in assessment of osteoporosis, equal to a patient's bone mineral density measurement by DEXA minus the value in a young healthy person, divided by the standard deviation of the measurement in the population.
  Participants
    Femoral total T-score ≤ -2.5 | 20 | 25 | 45
    Not Applicable | 153 | 145 | 298
T-score classification by inclusion criteria: Spine (average of spine Lumbar 1-4 ) T-score ≤-2.5 [Number; unit: Participants] — T-score: a measurement expressed in standard deviation units from a given mean used in assessment of osteoporosis, equal to a patient's bone mineral density measurement by DEXA minus the value in a young healthy person, divided by the standard deviation of the measurement in the population.
  Participants
    Spine (average of spine Lumbar 1-4 ) T-score ≤-2.5 | 144 | 132 | 276
    Not Applicable | 29 | 38 | 67
Two or more fractures in spine (Lumbar 1-4) [Number; unit: Participants]
  Two or more fractures in spine(Lumbar 1-4) | 3 | 4 | 7
  Not Applicable | 170 | 166 | 336
A fracture in spine Lumbar 1, Lumbar 2, Lumbar 3, Lumbar 4 and T-score ≤-2.0 [Mean (Standard Deviation); unit: T-score] — The analyzable number of patients with A fracture in spine Lumbar 1, Lumbar 2, Lumbar 3, Lumbar 4 and T-score ≤ -2.0 are 9 in Fosamax Plus D Group and 5 in Fosamax Group.
  T-score | -2.44 (0.71) | -2.34 (0.3) | -2.40 (0.59)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — 1 Participant from the Fosamax group is missing data for this Measure
  mm Hg | 72.5 (8.84) | 73.82 (8.85) | 73.15 (8.86)
Femoral neck T-score ≤ -2.5 [Mean (Standard Deviation); unit: T-score] — The analyzable number of patients with Femoral neck T-score ≤ -2.5 are 43 in Fosamax Plus D Group and 58 in Fosamax Group.
  T-score | -2.95 (0.48) | -2.94 (0.42) | -2.94 (0.45)
Femoral total T-score ≤ -2.5 [Mean (Standard Deviation); unit: T-score] — The analyzable number of patients with Femoral total T-score ≤ -2.5 are 20 in Fosamax Plus D Group and 25 in Fosamax Group.
  T-score | -3.00 (0.52) | -3.00 (0.41) | -3.00 (0.46)
Height [Mean (Standard Deviation); unit: Centimeters] — 2 Participants from the Fosamax group are missing data for this Measure
  Centimeters | 152.11 (5.88) | 152.47 (5.59) | 152.29 (5.73)
Serum PTH (Parathyroid hormone) [Mean (Standard Deviation); unit: pg/ml] | 25.27 (11.01) | 23.47 (11.85) | 24.38 (11.45)
Spine (average of spine Lumbar 1, Lumbar 2, Lumbar 3, Lumbar 4 ) T-score ≤ -2.5 [Mean (Standard Deviation); unit: T-score] — The analyzable number of patients with Spine (average of spine Lumbar 1, Lumbar 2, Lumbar 3, Lumbar 4) are 144 in Fosamax Plus D Group and 132 in Fosamax Group.
  T-score | -2.96 (0.40) | -3.06 (0.50) | -3.01 (0.45)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — 1 Participant from the Fosamax group is missing data for this Measure
  mm Hg | 122.83 (15.8) | 124.08 (14.52) | 123.45 (15.17)
Weight [Mean (Standard Deviation); unit: Kilograms] — 1 Participant from the Fosamax plus D group is missing data for this Measure, 2 Participants from the Fosamax group are missing data for this Measure
  Kilograms | 53.84 (6.89) | 54.8 (7.03) | 54.32 (6.97)
serum 25 OHD (Serum 25-hydroxyvitamin D) [Mean (Standard Deviation); unit: ng/ml] | 18.82 (6.46) | 18.71 (6.25) | 18.77 (6.35)

OUTCOME MEASURES:

1. Primary Outcome: Patients With Serum 25 OHD (Serum 25-hydroxyvitamin D) Below the Deficiency Level (Less Than 15 ng/ml) at 16 Weeks of Treatment
Time Frame: 16 weeks
Population: Participants for analysis was modified intention to treat (Number of patients : Fosamax Plus D Group was 136, Fosamax was 132). Missing data were imputed by the last observation carried forward (LOCF) technique.
Measure: Number; unit: participants
Groups:
- Fosamax Plus D: Once weekly Fosamax plus D tablet [Alendronate sodium 70 mg/Cholecalciferol 5600 IU] + once daily calcium formulation [500 mg/day]), 16 weeks and patients who 1) received at least one dose of investigational product, 2) performed efficacy assessment including pre-treatment value and at least one post-treatment value, 3) did not have any major protocol violations including enrollment prior to contract and the violation of drug administration and entry criteria
- Fosamax: Once weekly Fosamax 70 mg tablet [Alendronate sodium 70 mg] + once daily calcium formulation [500 mg/day], 16 weeks and patients who 1) received at least one dose of investigational product, 2) performed efficacy assessment including pre-treatment value and at least one post-treatment value, 3) did not have any major protocol violations including enrollment prior to contract and the violation of drug administration and entry criteria
Arm/Group | Fosamax Plus D | Fosamax
Number analyzed (Participants) | 136 | 132
participants
  With Vitamin D Deficiency | 2 | 55
  Without Vitamin D Deficiency | 134 | 77
Statistical Analysis 1: Comparison: Fosamax Plus D vs Fosamax; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Primary efficacy endpoint was analyzed by a Cochran-Mantel-Haenszel test with baseline vitamin D level as covariate; Odds Ratio (OR) = 0.02, 95% CI [0.00 to 0.08] — Mantel-Haenszel estimator of the common odds ratio was calculated by using Cochran-Mantel-Haenszel test for subjects' proportions with vitamin D deficiency changes at 16 weeks (visit 4) from baseline (visit 1) between treatment groups

2. Secondary Outcome: Serum PTH (Parathyroid Hormone) Percentage Changes From Baseline to 16 Weeks of Treatment
Time Frame: Baseline and 16 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change Serum PTH
Arm/Group | Fosamax Plus D | Fosamax
Number analyzed (Participants) | 136 | 132
Percentage Change Serum PTH | 8.17 [-3.24 to 19.58] | 29.98 [18.34 to 41.62]
Statistical Analysis 1: Comparison: Fosamax Plus D vs Fosamax; Test type: Superiority or Other; p = 0.0091, ANCOVA; Least squares mean is mean of serum PTH percentage changes adjusted serum PTH level at baseline

3. Post Hoc Outcome: Patients With Serum 25 OHD (Serum 25-hydroxyvitamin D) Less and Greater Than 20 ng/ml at 16 Weeks of Treatment
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Fosamax Plus D | Fosamax
Number analyzed (Participants) | 136 | 132
participants
  With 25 OHD < 20ng/ml at 16 weeks of treatment | 7 | 93
  With 25 OHD >= 20ng/ml at 16 weeks of treatment | 129 | 39
Statistical Analysis 1: Comparison: Fosamax Plus D vs Fosamax; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; It was analyzed by a Cochran-Mantel-Haenszel test with baseline vitamin D level as covariate; Odds Ratio (OR) = 0.02, 95% CI [0.01 to 0.04] — [estimate comment as in outcome 1, analysis 1]

4. Post Hoc Outcome: Mean Serum 25 OHD(Serum 25-hydroxyvitamin D) at 16 Weeks of Treatment
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Fosamax Plus D | Fosamax
Number analyzed (Participants) | 136 | 132
ng/ml | 30.08 (5.87) | 17.14 (6.04)

ADVERSE EVENTS:
Time Frame: Adverse events were followed up until 14 days after the last dose of investigational drug.
Description: 1 Participant from Fosamax Plus D Group and 1 participant from Fosamax Group were not actually administered study drug after randomization and were exclude in AE reporting Group.
  1 participant from Fosamax Plus D group was actually administered Fosamax and analyzed as Fosamax Group in AE reporting Group.
Groups:
- Fosamax Plus D: Once weekly Fosamax plus D tablet [Alendronate sodium 70 mg/Cholecalciferol 5600 IU] + once daily calcium formulation [500 mg/day]), 16 weeks and patients who received drugs at least once after randomization and was analyzed according to the actually administered study drugs
- Fosamax: Once weekly Fosamax 70 mg tablet [Alendronate sodium 70 mg] + once daily calcium formulation [500 mg/day]), 16 weeks and patients who received drugs at least once after randomization and was analyzed according to the actually administered study drugs
Arm/Group | Fosamax Plus D | Fosamax
Serious Adverse Events (participants affected / at risk) | 7/171 | 1/170
Other Adverse Events (participants affected / at risk) | 60/171 | 55/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosamax Plus D (N=171) | Fosamax (N=170)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosamax Plus D (N=171) | Fosamax (N=170)
Dyspepsia (Gastrointestinal disorders) | 11 (11) | 18 (18)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (12) | 8 (9)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Asthenia (General disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 2 (2)
Chills (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.